CLINICAL TRIAL: NCT03277313
Title: Efficacy, Safety, Tolerability, Immunogenicity and Pharmacokinetic Evaluation of HYQVIA in Pediatric Subjects With Primary Immunodeficiency Diseases
Brief Title: Efficacy, Safety, Tolerability, Immunogenicity and Pharmacokinetic Evaluation of HYQVIA in Pediatric PIDD Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 161503
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Epoch 1 (Experimental): Pediatric participants with PIDD who were on IV or non-HYQVIA SC treatment with immunoglobulin were enrolled and treated with HYQVIA SC with a dose or interval ramp-up period of up to six weeks. HYQVIA dose was planned to be equivalent to 100% (± 5%) of pre-study treatment. Dose frequency was one treatment interval of one week, then one treatment interval of two weeks for participants who were planned to be treated every three weeks, and one more treatment interval of three weeks for participants who were planned to be treated every four weeks.
  Interventions: Biological: HYQVIA
- Epoch 2 (Experimental): Epoch 1 was followed by Epoch 2 with HYQVIA treatment infusions given once every 3 or 4 weeks, depending on the participant's previous IV dosing schedule (for IV pretreated participants) and at the discretion of the investigator and participant (for SC-pretreated participants) up to approximately 36 months.
  Interventions: Biological: HYQVIA

INTERVENTIONS:
Biological: HYQVIA — Immune Globulin Infusion 10% (Human) with Recombinant Human Hyaluronidase (IGI, 10% with rHuPH20)
  Other Names: IGI 10% with rHuPH20

SUMMARY:
The purpose of the study is to acquire additional data on efficacy, safety, tolerability, immunogenicity, pharmacokinetic (PK) and other parameters of HYQVIA in pediatric (age ≥ 2 to <16 years) participants with primary immunodeficiency disease (PIDD).

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have a documented diagnosis of a form of primary immunodeficiency (PI) involving a defect in antibody formation and requiring gammaglobulin replacement, as defined according to the International Union of Immunological Societies (IUIS) Scientific Committee 2015 (Picard et al., 2015) prior to enrollment. The diagnosis must be confirmed by the sponsor´s Medical Director prior to first treatment with IP in the study.
2. Participant is at least two and below 16 years of age at the time of screening.
3. Participant has been receiving a consistent dose of Immunoglobulin G (IgG), administered in compliance with the respective product information for a period of at least three months prior to screening. The average minimum pre-study dose over that interval was equivalent to 300 mg/kg BW / 4 weeks and a maximum dose equivalent to 1000 mg/kg body weight (BW) / 4 weeks.
4. Participant has a serum trough level of IgG > 5 g/L at screening.
5. If female of childbearing potential, participant presents with a negative pregnancy test and agrees to employ adequate birth control measures for the duration of the study.
6. Participant /legally authorized representative is willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Participant has a known history of or is positive at screening for one or more of the following: hepatitis B surface antigen (HBsAg), polymerase chain reaction (PCR) for hepatitis C virus (HCV), PCR for human immunodeficiency virus (HIV) Type 1/2.
2. Abnormal laboratory values at screening meeting any one of the following criteria (abnormal tests may be repeated once to determine if they are persistent):

   1. Persistent alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 times the upper limit of normal (ULN) for the testing laboratory
   2. Persistent severe neutropenia (defined as an absolute neutrophil count [ANC] ≤ 500/mm^3)
3. Participant has anemia that would preclude phlebotomy for laboratory studies, according to standard practice at the site.
4. Participant has an ongoing history of hypersensitivity or persistent reactions (urticaria, breathing difficulty, severe hypotension, or anaphylaxis) following intravenous (IV) immunoglobulin, subcutaneous (SC) immunoglobulin, and/or Immune Serum Globulin (ISG) infusions.
5. Participant has severe Immunoglobulin A (IgA) deficiency (less than 7.0 mg/dL) with known anti-IgA antibodies and a history of hypersensitivity.
6. Participant has a known allergy to hyaluronidase.
7. Participant has active infection and is receiving antibiotic therapy for the treatment of infection at the time of screening.
8. Participant has a bleeding disorder or a platelet count less than 20,000/μL, or who, in the opinion of the investigator, would be at significant risk of increased bleeding or bruising as a result of SC therapy.
9. Participant has severe dermatitis that would preclude adequate sites for safe product administration in the opinion of the investigator.
10. Participant has participated in another clinical study involving an IP or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
11. Participant is a family member or employee of the investigator.
12. If female, participant is pregnant or lactating at the time of enrollment.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (19):
- United States (19):
  - University of Alabama Medical Center, Birmingham, Alabama
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - University of Miami Pediatric Allergy and Immunology, Miami, Florida
  - University of South Florida Physician Group, St. Petersburg, Florida
  - Georgia Pollens Clinical Research Centers, Inc., Albany, Georgia
  - Emory Healthcare, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Women & Children's Hospital of Buffalo, Buffalo, New York
  - Northwell Health, Inc. PRIME, Great Neck, New York
  - Stony Brook Children's Hospital, Stony Brook, New York
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Allergy Asthma & Immunology Relief of Charlotte, Charlotte, North Carolina
  - OK Institute of Allergy & Asthma Clinical Research, LLC, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Allergy Partners of North Texas Research, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Section on Immunopathogenesis and Clinical Immunology, Fairfax, Virginia
  - Marshall University Joan C. Edwards School of Medicine, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc54db2bf003ab45c6c

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 19 investigative sites in the United States from 25 September 2017 to 20 July 2022. Pediatric participants with a diagnosis of primary immunodeficiency diseases (PIDD) were enrolled in this study.
Pre-assignment Details: Pediatric participants who received intravenous(IV) or non-HYQVIA subcutaneous(SC) immunoglobulin therapy prior to enrollment received ramp-up doses of HYQVIA in Epoch 1 and at 3- or 4-week intervals in Epoch 2. Epoch 3 was planned for safety follow-up if needed, however no participants continued in Epoch 3. Data is reported only for Epoch 1 and 2.
Period: Epoch 1 (Six-week Ramp-up Period)
Arm/Group | Epoch 1 | Epoch 2
Started | 44 | 0
Completed | 43 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Epoch 2 (36 Months After Epoch 1)
Arm/Group | Epoch 1 | Epoch 2
Started | 0 | 43
Completed | 0 | 34
Not Completed | 0 | 9
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 6
Not completed — Reason not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who provided informed consent, and met enrollment eligibility.
Arm/Group | Epoch 1
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (3.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 40
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44
Height [Mean (Standard Deviation); unit: cm] | 133.60 (24.024)
Weight [Mean (Standard Deviation); unit: kg] | 37.78 (19.858)

OUTCOME MEASURES:

1. Primary Outcome: Rate Represented as Mean Number of Acute Serious Bacterial Infections (ASBI) Per Participant-year
Description: The rate of ASBI was defined as the mean number of ASBI per participant-year based on the United States (U.S.) Food and drugs Administration (FDA) guidance for industry to support marketing of human immune globulin intravenous (IGIV) as replacement therapy for primary humoral immunodeficiency and the European Medicines Agency (EMA) guideline on the clinical investigation of human normal immunoglobulin for SC and /or intramuscular administration. ASBI included bacteremia/sepsis, bacterial meningitis, osteomyelitis/septic arthritis, bacterial pneumonia, and visceral abscess, diagnosed according to the Diagnostic Criteria for Acute Serious Bacterial Infections.
Time Frame: From first dose of study drug up to end of Study Epoch 2 (up to approximately 37.2 months)
Population: FAS included all participants who provided informed consent, and met enrollment eligibility.
Measure: Mean (Standard Error); unit: ASBI per participant-year
Groups:
- Epoch 1 + Epoch 2: Pediatric participants with PIDD who were on IV or non-HYQVIA SC treatment with immunoglobulin were enrolled and treated with HYQVIA SC with a dose or interval ramp-up period of up to six weeks. HYQVIA dose was planned to be equivalent to 100% (± 5%) of pre-study treatment. Dose frequency was one treatment interval of one week, then one treatment interval of two weeks for participants who were planned to be treated every three weeks, and one more treatment interval of three weeks for participants who were planned to be treated every four weeks. Epoch 1 was followed by Epoch 2 with HYQVIA treatment infusions given once every 3 or 4 weeks, depending on the participant's previous IV dosing schedule (for IV pretreated participants) and at the discretion of the investigator and participant (for SC-pretreated participants) up to approximately 36 months.
Arm/Group | Epoch 1 + Epoch 2
Number analyzed (Participants) | 44
ASBI per participant-year | 0.04 (0.027)

2. Secondary Outcome: Rate Represented as Mean Number of All Infections Per Participant-year
Description: The rate of all infections was defined as the mean number of all infections per participant-year. Number of all infections was calculated as number of infections per participant-year.
Time Frame: From first dose of study drug up to end of Study Epoch 2 (up to approximately 37.2 months)
Population: FAS included all participants who provided informed consent, and met enrollment eligibility.
Measure: Mean (Standard Error); unit: infections per participant-year
Arm/Group | Epoch 1 + Epoch 2
Number analyzed (Participants) | 44
infections per participant-year | 3.12 (0.450)

3. Secondary Outcome: Epoch 2: Trough Levels of Immunoglobulin G (IgG) Total and IgG Subclasses
Time Frame: Study Epoch 2, Year 1: Months 0, 6, and 12; Year 2: Months 18, 24 and 36
Population: FAS=all participants who provided informed consent, and met enrollment eligibility. Only FAS participants in Epoch 2 were analyzed for this outcome measure. Overall number analyzed=number of participants with data available for analyses. Number analyzed=number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Epoch 2
Number analyzed (Participants) | 40
grams per liter (g/L)
  IgG Total: Month 0 | 10.381 (2.9191)
  IgG Total: Month 6: number analyzed (Participants) | 33
  IgG Total: Month 6 | 9.199 (1.9577)
  IgG Total: Month 12: number analyzed (Participants) | 36
  IgG Total: Month 12 | 9.214 (1.9800)
  IgG Total: Month 18: number analyzed (Participants) | 1
  IgG Total: Month 18 | 13.80 (NA) — Standard deviation (SD) was not estimable for 1 participant.
  IgG Total: Month 24: number analyzed (Participants) | 1
  IgG Total: Month 24 | 10.80 (NA) — SD was not estimable for 1 participant.
  IgG Total: Month 36: number analyzed (Participants) | 1
  IgG Total: Month 36 | 13.50 (NA) — SD was not estimable for 1 participant.
  IgG Subclass 1: Month 0: number analyzed (Participants) | 39
  IgG Subclass 1: Month 0 | 5.888 (2.7193)
  IgG Subclass 1: Month 6: number analyzed (Participants) | 39
  IgG Subclass 1: Month 6 | 5.317 (1.4887)
  IgG Subclass 1: Month 12: number analyzed (Participants) | 36
  IgG Subclass 1: Month 12 | 5.284 (1.2103)
  IgG Subclass 1: Month 18: number analyzed (Participants) | 1
  IgG Subclass 1: Month 18 | 7.590 (NA) — SD was not estimable for 1 participant.
  IgG Subclass 1: Month 24: number analyzed (Participants) | 1
  IgG Subclass 1: Month 24 | 7.710 (NA) — SD was not estimable for 1 participant.
  IgG Subclass 1: Month 36: number analyzed (Participants) | 0
  IgG Subclass 2: Month 0: number analyzed (Participants) | 39
  IgG Subclass 2: Month 0 | 3.311 (0.6833)
  IgG Subclass 2: Month 6: number analyzed (Participants) | 39
  IgG Subclass 2: Month 6 | 3.156 (0.6694)
  IgG Subclass 2: Month 12: number analyzed (Participants) | 36
  IgG Subclass 2: Month 12 | 3.106 (0.5839)
  IgG Subclass 2: Month 18: number analyzed (Participants) | 1
  IgG Subclass 2: Month 18 | 3.480 (NA) — SD was not estimable for 1 participant.
  IgG Subclass 2: Month 24: number analyzed (Participants) | 1
  IgG Subclass 2: Month 24 | 3.510 (NA) — SD was not estimable for 1 participant.
  IgG Subclass 2: Month 36: number analyzed (Participants) | 0
  IgG Subclass 3: Month 0: number analyzed (Participants) | 39
  IgG Subclass 3: Month 0 | 0.534 (0.2838)
  IgG Subclass 3: Month 6: number analyzed (Participants) | 39
  IgG Subclass 3: Month 6 | 0.508 (0.2545)
  IgG Subclass 3: Month 12: number analyzed (Participants) | 36
  IgG Subclass 3: Month 12 | 0.507 (0.2799)
  IgG Subclass 3: Month 18: number analyzed (Participants) | 1
  IgG Subclass 3: Month 18 | 0.360 (NA) — SD was not estimable for 1 participant.
  IgG Subclass 3: Month 24: number analyzed (Participants) | 1
  IgG Subclass 3: Month 24 | 0.430 (NA) — SD was not estimable for 1 participant.
  IgG Subclass 3: Month 36: number analyzed (Participants) | 0
  IgG Subclass 4: Month 0: number analyzed (Participants) | 39
  IgG Subclass 4: Month 0 | 0.2998 (0.26802)
  IgG Subclass 4: Month 6: number analyzed (Participants) | 39
  IgG Subclass 4: Month 6 | 0.3161 (0.32899)
  IgG Subclass 4: Month 12: number analyzed (Participants) | 36
  IgG Subclass 4: Month 12 | 0.3118 (0.32790)
  IgG Subclass 4: Month 18: number analyzed (Participants) | 1
  IgG Subclass 4: Month 18 | 0.9380 (NA) — SD was not estimable for 1 participant.
  IgG Subclass 4: Month 24: number analyzed (Participants) | 1
  IgG Subclass 4: Month 24 | 1.4560 (NA) — SD was not estimable for 1 participant.
  IgG Subclass 4: Month 36: number analyzed (Participants) | 0

4. Secondary Outcome: Epoch 2: Trough Levels of Specific Antibodies to Clinically Relevant Pathogens Categorized as Clostridium Tetani Toxoid and Hepatitis B Virus
Time Frame: Study Epoch 2, Year 2: Months 6, 24, and 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: international unit per milliliter(IU/mL)
Arm/Group | Epoch 2
Number analyzed (Participants) | 38
international unit per milliliter(IU/mL)
  Clostridium Tetani Toxoid Antibody: Month 6: number analyzed (Participants) | 36
  Clostridium Tetani Toxoid Antibody: Month 6 | 1.685 (0.6793)
  Clostridium Tetani Toxoid Antibody: Month 24: number analyzed (Participants) | 1
  Clostridium Tetani Toxoid Antibody: Month 24 | 2.450 (NA) — SD was not estimable for one participant.
  Clostridium Tetani Toxoid Antibody: Completion/ Termination (Month 36): number analyzed (Participants) | 37
  Clostridium Tetani Toxoid Antibody: Completion/ Termination (Month 36) | 1.598 (0.5889)
  Hepatitis B Virus Antibody: Month 6: number analyzed (Participants) | 36
  Hepatitis B Virus Antibody: Month 6 | 199.6 (122.97)
  Hepatitis B Virus Antibody: Month 24: number analyzed (Participants) | 1
  Hepatitis B Virus Antibody: Month 24 | 146.0 (NA) — SD was not estimable for 1 participant.
  Hepatitis B Virus Antibody: Completion/ Termination (Month 36) | 256.7 (219.53)

5. Secondary Outcome: Epoch 2: Trough Levels of Specific Antibodies to Clinically Relevant Pathogen Haemophilus Influenzae B
Time Frame: Study Epoch 2, Year 2: Months 6, 24, and 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Epoch 2
Number analyzed (Participants) | 39
milligrams per liter (mg/L)
  Month 6: number analyzed (Participants) | 36
  Month 6 | 1.839 (1.5222)
  Month 24: number analyzed (Participants) | 1
  Month 24 | 1.810 (NA) — SD was not estimable for 1 participant.
  Completion/Termination (Month 36) | 1.678 (0.8009)

6. Secondary Outcome: Epoch 2: Area Under the Curve Normalized for Week (AUCweek)
Time Frame: Study Epoch 2, Month 6: Day 0 pre-infusion, and at Days 2, 4, 10, 21 and 28 post-infusion
Population: Pharmacokinetic analysis set (PKAS) included all participants in the Safety Analysis Set who have at least 1 evaluable post-dose concentration data for PK assessments without major protocol deviations or events affecting the PK results. Overall number analyzed is the number of participants with data available for analyses. As pre-specified in statistical analysis plan (SAP), this outcome measure was planned only for Epoch 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: grams*day per liter (g*day/L)
Arm/Group | Epoch 2
Number analyzed (Participants) | 37
grams*day per liter (g*day/L) | 74.57 (19.4)

7. Secondary Outcome: Epoch 2: Area Under the Curve Over the Infusion Interval (AUCTau)
Time Frame: Study Epoch 2, Month 6: Day 0 pre-infusion, and at Days 2, 4, 10, 21 and 28 post-infusion
Population: PKAS included all participants in the Safety Analysis Set who have at least 1 evaluable post-dose concentration data for PK assessments without major protocol deviations or events affecting the PK results. Overall number analyzed is the number of participants with data available for analyses. As pre-specified in SAP, this outcome measure was planned only for Epoch 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: g*day/L
Arm/Group | Epoch 2
Number analyzed (Participants) | 37
g*day/L | 288.8 (21.7)

8. Secondary Outcome: Epoch 2: Apparent Clearance (CL/F)
Time Frame: Study Epoch 2, Month 6: Day 0 pre-infusion, and at Days 2, 4, 10, 21 and 28 post-infusion
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per day (mL/day)
Arm/Group | Epoch 2
Number analyzed (Participants) | 37
milliliters per day (mL/day) | 56.45 (61.4)

9. Secondary Outcome: Epoch 2: Maximum Concentration (Cmax)
Time Frame: Study Epoch 2, Month 6: Day 0 pre-infusion, and at Days 2, 4, 10, 21 and 28 post-infusion
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: g/L
Arm/Group | Epoch 2
Number analyzed (Participants) | 38
g/L | 12.94 (17.4)

10. Secondary Outcome: Epoch 2: Minimum Concentration (Cmin)
Time Frame: Study Epoch 2, Month 6: Day 0 pre-infusion, and at Days 2, 4, 10, 21 and 28 post-infusion
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: g/L
Arm/Group | Epoch 2
Number analyzed (Participants) | 38
g/L | 8.571 (25.6)

11. Secondary Outcome: Epoch 2: Time to Maximum Concentration (Tmax)
Time Frame: Study Epoch 2, Month 6: Day 0 pre-infusion, and at Days 2, 4, 10, 21 and 28 post-infusion
Population: as for outcome 7
Measure: Median (Full Range); unit: days
Arm/Group | Epoch 2
Number analyzed (Participants) | 38
days | 4.20 [0.0 to 26.9]

12. Secondary Outcome: Epoch 2: Terminal Half-life (T 1/2)
Time Frame: Study Epoch 2, Month 6: Day 0 pre-infusion, and at Days 2, 4, 10, 21 and 28 post-infusion
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Epoch 2
Number analyzed (Participants) | 19
days | 44.98 (45.9)

13. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) Excluding Infections, Related and Not Related
Description: An SAE is defined as an untoward medical occurrence that at any dose is fatal, life-threatening, requires inpatient hospitalization or results in prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event. Number of participants who experienced SAEs, related or not related, was reported.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: Safety Analysis Set (SAS) included all participants who received at least one dose of HyQvia.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1 | Epoch 2
Number analyzed (Participants) | 44 | 43
Participants
  SAE: Related | 0 | 0
  SAE: Not Related | 0 | 1

14. Secondary Outcome: Rate of SAEs Excluding Infections, Related and Not Related, Per Infusion
Description: Rate of SAEs per infusion was calculated as number of serious adverse events/total number of infusions administered to participants in the analysis set. Rate of SAEs per infusion (excluding infections) was reported.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Number; unit: SAEs per infusion
Units Other Than Participants: Infusions
Arm/Group | Epoch 1 | Epoch 2
Number analyzed (Participants) | 44 | 43
Number analyzed (Infusions) | 126 | 633
SAEs per infusion
  SAE: Related | 0.0 | 0.0
  SAE: Not Related | 0.0 | 0.002

15. Secondary Outcome: Number of Participants With All Treatment Emergent Adverse Events (TEAEs) Excluding Infections, Related and Not Related
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. Number of participants who experienced TEAEs, related or not related, was reported.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1 | Epoch 2
Number analyzed (Participants) | 44 | 43
Participants
  TEAE: Related | 25 | 31
  TEAE: Not Related | 16 | 36

16. Secondary Outcome: Rate of All TEAEs Excluding Infections, Related and Not Related, Per Infusion
Description: Rate of all TEAEs per infusion was calculated as number of any adverse reaction events/total number of infusions administered to participants in the analysis set. Rate of any adverse reactions per infusion (excluding infections) was reported.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Number; unit: adverse reaction event per infusion
Units Other Than Participants: Infusion
Arm/Group | Epoch 1 | Epoch 2
Number analyzed (Participants) | 44 | 43
Number analyzed (Infusion) | 126 | 633
adverse reaction event per infusion
  TEAE: Related | 0.675 | 0.397
  TEAE: Not Related | 0.270 | 0.262

17. Secondary Outcome: Number of Participants With Local TEAEs Excluding Infections, Related and Not Related
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. Number of participants who experienced local TEAEs, related or not related, was reported.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1 | Epoch 2
Number analyzed (Participants) | 44 | 43
Participants
  Local TEAE: Related | 22 | 28
  Local TEAE: Not Related | 2 | 6

18. Secondary Outcome: Rate of Local TEAEs Excluding Infections, Related and Not Related, Per Infusion
Description: Rate of local TEAEs per infusion was calculated as number of local TEAEs/total number of infusions administered to participants in the analysis set. Rate of local TEAEs per infusion (excluding infections) was reported.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Number; unit: local TEAEs per infusion
Units Other Than Participants: Infusion
Arm/Group | Epoch 1 | Epoch 2
Number analyzed (Participants) | 44 | 43
Number analyzed (Infusion) | 126 | 633
local TEAEs per infusion
  Local TEAE: Related | 0.460 | 0.212
  Local TEAE: Not Related | 0.016 | 0.013

19. Secondary Outcome: Number of Participants With Systemic TEAEs Excluding Infections, Related and Not Related
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. Number of participants who experienced systemic TEAEs, related or not related, was reported.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1 | Epoch 2
Number analyzed (Participants) | 44 | 43
Participants
  Systemic TEAE: Related | 12 | 20
  Systemic TEAE: Not Related | 16 | 33

20. Secondary Outcome: Rate of Systemic TEAEs Excluding Infections, Related and Not Related, Per Infusion
Description: Rate of systemic TEAEs per infusion was calculated as number of systemic TEAEs/total number of infusions administered to participants in the analysis set. Rate of systemic TEAEs per infusion (excluding infections) was reported.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Number; unit: systemic TEAEs per infusion
Units Other Than Participants: Infusion
Arm/Group | Epoch 1 | Epoch 2
Number analyzed (Participants) | 44 | 43
Number analyzed (Infusion) | 126 | 633
systemic TEAEs per infusion
  Systemic TEAE: Related | 0.214 | 0.185
  Systemic TEAE: Not Related | 0.254 | 0.250

21. Secondary Outcome: Number of Participants With All Temporally Associated TEAEs Excluding Infections
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. TEAE is defined as an adverse event with an onset that occurs after receiving study drug. Number of participants who experienced all temporally associated TEAEs, related or not related, was reported.
Time Frame: From beginning of infusion up to 72 hours post infusion
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1 | Epoch 2
Number analyzed (Participants) | 44 | 43
Participants | 27 | 35

22. Secondary Outcome: Rate of All Temporally Associated TEAEs Excluding Infections Per Infusion
Description: Rate of all temporally associated TEAEs per infusion was calculated as number of all temporally associated TEAEs/total number of infusions administered to participants in the analysis set. Rate of all temporally associated TEAEs per infusion (excluding infections) was reported.
Time Frame: From beginning of infusion up to 72 hours post infusion
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Number; unit: temporally associated TEAEs per infusion
Units Other Than Participants: Infusion
Arm/Group | Epoch 1 | Epoch 2
Number analyzed (Participants) | 44 | 43
Number analyzed (Infusion) | 126 | 633
temporally associated TEAEs per infusion | 0.722 | 0.460

23. Secondary Outcome: Number of Participants With All Related (Causally) and/or Temporally Associated TEAEs Excluding Infections
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. Number of participants with any related (causally) and/or temporally associated TEAEs (excluding infections) was reported. Temporally-associated TEAEs were defined as TEAEs which begin during infusion of IP or within 72 hours following the end of IP infusion.
Time Frame: From beginning of infusion up to 72 hours post infusion
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1 | Epoch 2
Number analyzed (Participants) | 44 | 43
Participants | 27 | 35

24. Secondary Outcome: Rate of Participants With All Related (Causally) and/or Temporally Associated TEAEs Excluding Infections Per Infusion
Description: Rate of any related (causally) and/or temporally associated TEAEs per infusion was calculated as number of related and/or temporally associated adverse events/ total number of infusions administered to participants in the analysis set. TEAEs recorded in the study database as "possibly related" or "probably related" to HYQVIA are considered HYQVIA-related adverse events. Temporally-associated TEAEs were defined as TEAEs which begin during infusion of IP or within 72 hours following the end of IP infusion. Rate of any related (causally) and/or temporally associated TEAEs per infusion (excluding infections) was reported.
Time Frame: From beginning of infusion up to 72 hours post infusion
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Number; unit: related temporally TEAEs per infusion
Units Other Than Participants: Infusion
Arm/Group | Epoch 1 | Epoch 2
Number analyzed (Participants) | 44 | 43
Number analyzed (Infusion) | 126 | 633
related temporally TEAEs per infusion | 0.762 | 0.482

25. Secondary Outcome: Percentage of Participants With Any TEAEs Excluding Infections
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 1 | Epoch 2
Number analyzed (Participants) | 44 | 43
percentage of participants | 65.9 | 93.0

26. Secondary Outcome: Number of Participants Who Developed Positive Titer (≥160) of Binding or Neutralizing Antibodies to rHuPH20
Description: Number of participants who developed positive titer (rHuPH20 titer ≥160) of binding antibodies to rHuPH20 was reported. Neutralizing antibodies were only tested if the participant had a titer of ≥160 of binding antibodies. Participants with multiple assessments of titer of ≥160 of binding antibodies are counted only once.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: FAS included all participants who provided informed consent, and met enrollment eligibility.
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 1 + Epoch 2
Number analyzed (Participants) | 44
Participants | 1

27. Secondary Outcome: Percentage of Participants Who Developed Positive Titer (≥160) of Binding or Neutralizing Antibodies to rHuPH20
Description: Percentage of participants who developed positive titer (rHuPH20 titer ≥160) of binding antibodies to rHuPH20 was reported. Neutralizing antibodies were only tested if the participant had a titer of ≥160 of binding antibodies. Participants with multiple assessments of titer of ≥160 of binding antibodies are counted only once. Percentages are rounded off to whole number at the nearest decimal.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: FAS included all participants who provided informed consent, and met enrollment eligibility.
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 1 + Epoch 2
Number analyzed (Participants) | 44
percentage of participants | 2.3

28. Secondary Outcome: Epoch 2: Number of Infusions Per Month
Time Frame: Study Epoch 2: Up to 36 months
Population: SAS included all participants who received at least one dose of HyQvia. As pre-specified in SAP, this outcome measure was planned only for Epoch 2.
Measure: Median (Full Range); unit: infusions per month
Arm/Group | Epoch 2
Number analyzed (Participants) | 43
infusions per month | 1.10 [1.0 to 1.5]

29. Secondary Outcome: Epoch 2: Number of Infusion Sites (Needle Sticks) Per Infusion
Time Frame: Study Epoch 2: Up to 36 months
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: infusion sites per infusion
Units Other Than Participants: Infusion
Arm/Group | Epoch 2
Number analyzed (Participants) | 43
Number analyzed (Infusion) | 633
infusion sites per infusion | 1.83 (0.366)

30. Secondary Outcome: Epoch 2: Number of Infusion Sites (Needle Sticks) Per Month
Time Frame: Study Epoch 2: Up to 36 months
Population: as for outcome 28
Measure: Median (Full Range); unit: infusion sites per month
Arm/Group | Epoch 2
Number analyzed (Participants) | 43
infusion sites per month | 2.17 [1.1 to 2.9]

31. Secondary Outcome: Epoch 2: Duration of Infusion
Description: Duration of infusion is calculated as (stop time of infusion - start time of infusion) (in Epoch 2). Duration of infusion is the time from the start of rHuPH20 infusion until the stop time of immunoglobulin infusion.
Time Frame: Study Epoch 2: Up to 36 months
Population: as for outcome 28
Measure: Median (Full Range); unit: minutes (mins)
Units Other Than Participants: Infusion
Arm/Group | Epoch 2
Number analyzed (Participants) | 43
Number analyzed (Infusion) | 632
minutes (mins) | 85.0 [45 to 215]

32. Secondary Outcome: Epoch 2: Maximum Infusion Rate Per Site
Description: HYQVIA treatment infusions in Epoch 2 were given at a rate of 10 milliliters per hour per site (mL/h/site) to 160 ml/h/site (body weight [BW] of <40 kg) and 10 mL/h/site to 300 mL/h/site (BW of ≥40 kg).
Time Frame: Study Epoch 2: Up to 36 months
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: milliliters per hour per site(mL/h/site)
Units Other Than Participants: Infusion
Arm/Group | Epoch 2
Number analyzed (Participants) | 43
Number analyzed (Infusion) | 633
milliliters per hour per site(mL/h/site) | 173.5 (81.32)

33. Secondary Outcome: Epoch 2: Infusion Volume Per Site
Description: Infusion volume per site is calculated as (actual IgG volume (mL) / total number of infusion sites used).
Time Frame: Study Epoch 2: Up to 36 months
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: mL/site
Units Other Than Participants: Infusion
Arm/Group | Epoch 2
Number analyzed (Participants) | 43
Number analyzed (Infusion) | 633
mL/site | 101.3 (51.69)

34. Secondary Outcome: Epoch 2: Infusions Which Were Discontinued, Slowed, or Interrupted Due to an AE
Time Frame: Study Epoch 2: Up to 36 months
Population: as for outcome 28
Measure: Number; unit: infusions
Units Other Than Participants: Infusion
Arm/Group | Epoch 2
Number analyzed (Participants) | 43
Number analyzed (Infusion) | 633
infusions
  Infusions That Were Discontinued | 0
  Infusions That Were Slowed | 0
  Infusions That Were Interrupted | 17

35. Secondary Outcome: Epoch 2: Percentage of Infusions Which Were Discontinued, Slowed, or Interrupted Due to an AE
Description: Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Study Epoch 2: Up to 36 months
Population: as for outcome 28
Measure: Number; unit: percentage of infusions
Units Other Than Participants: Infusion
Arm/Group | Epoch 2
Number analyzed (Participants) | 43
Number analyzed (Infusion) | 633
percentage of infusions
  Infusions That Were Discontinued | 0
  Infusions That Were Slowed | 0
  Infusions That Were Interrupted | 2.69

36. Secondary Outcome: Epoch 1: Number of Weeks to Reach Final Dose Interval
Time Frame: Epoch 1 (up to 6 weeks)
Population: SAS included all participants who received at least one dose of HyQvia. Overall number analyzed is the number of participants with data available for analyses. As pre-specified in SAP, this outcome measure was planned only for Epoch 1.
Measure: Median (Full Range); unit: weeks
Arm/Group | Epoch 1
Number analyzed (Participants) | 43
weeks | 6.14 [3.0 to 6.6]

37. Secondary Outcome: Epoch 2: Percentage of Participants Who Achieved a Treatment Interval of Three or Four Weeks in Epoch 2
Description: Percentages are rounded off to whole number at the nearest decimal. Percentages may sum up to more than 100% as assigned treatment interval could be changed during the study.
Time Frame: Study Epoch 2: Up to 36 months
Population: as for outcome 28
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 2
Number analyzed (Participants) | 43
percentage of participants
  Every 3 Weeks | 18.6
  Every 4 Weeks | 83.7

38. Secondary Outcome: Epoch 2: Percentage of Participants Who Maintained a Treatment Interval of Three or Four Weeks in Epoch 2 for 12 Months
Description: Percentages are rounded off to whole number at the nearest decimal.
Time Frame: Study Epoch 2: Up to 12 months
Population: as for outcome 28
Measure: Number; unit: percentage of participants
Arm/Group | Epoch 2
Number analyzed (Participants) | 43
percentage of participants | 74.4

39. Secondary Outcome: Health-related Quality of Life (HRQoL): Change From Baseline in Pediatric Quality of Life Inventory (Peds-QL) Score
Description: Peds-QL=generic questionnaire developed and validated to measure HRQoL among pediatric population. It included assessment of 4 dimensions: physical functioning (8 items), emotional functioning (8 items), social functioning (8 items), and school functioning (Age groups: Toddler (2-4years),Young child (5-7years),Child (8-12years), and Teens (13-<16years). Depending on the participants age, questionnaire may be completed by participant or parent/caregiver as appropriate. Items were scored on a 5-point Likert scale: 0=never a problem; 1=almost never a problem; 2=sometimes a problem; 3=often a problem; and 4=almost always a problem). All Scores were transformed on a total scale from 0-100 where, 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores indicating better health status. End of Epoch 2 summarizes all participant's data for their last epoch 2 visit (so not including the participant that discontinued in epoch 1).
Time Frame: Epoch 1: Baseline (First Infusion); Study Epoch 2: Up to Month 36
Population: SAS included all participants who received at least one dose of HyQvia. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at a specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epoch 1 + Epoch 2
Number analyzed (Participants) | 18
score on a scale
  Baseline: 2-4 years: number analyzed (Participants) | 8
  Baseline: 2-4 years | 72.67 (12.969)
  Baseline: 5-7 years: number analyzed (Participants) | 8
  Baseline: 5-7 years | 77.29 (18.908)
  Baseline: 8-12 years: number analyzed (Participants) | 8
  Baseline: 8-12 years | 75.42 (17.227)
  Baseline: 13-<16 years: number analyzed (Participants) | 8
  Baseline: 13-<16 years | 76.09 (7.894)
  Change From Baseline at Epoch 2 Month 12: 2-4 years: number analyzed (Participants) | 7
  Change From Baseline at Epoch 2 Month 12: 2-4 years | 4.57 (17.134)
  Change From Baseline at Epoch 2 Month 12: 5-7 years: number analyzed (Participants) | 9
  Change From Baseline at Epoch 2 Month 12: 5-7 years | -3.74 (15.170)
  Change From Baseline at Epoch 2 Month 12: 8-12 years: number analyzed (Participants) | 13
  Change From Baseline at Epoch 2 Month 12: 8-12 years | 0.84 (21.050)
  Change From Baseline at Epoch 2 Month 12: 13-<16 years: number analyzed (Participants) | 5
  Change From Baseline at Epoch 2 Month 12: 13-<16 years | -6.09 (8.750)
  Change From Baseline at Completion/ termination (Month 36): 2-4 years: number analyzed (Participants) | 3
  Change From Baseline at Completion/ termination (Month 36): 2-4 years | 8.73 (18.799)
  Change From Baseline at Completion/ termination (Month 36): 5-7 years: number analyzed (Participants) | 1
  Change From Baseline at Completion/ termination (Month 36): 5-7 years | -26.09 (NA) — SD was not estimable for 1 participant.
  Change From Baseline at Completion/ termination (Month 36): 8-12 years: number analyzed (Participants) | 8
  Change From Baseline at Completion/ termination (Month 36): 8-12 years | -5.16 (19.735)
  Change From Baseline at Completion/ termination (Month 36): 13-<16 years: number analyzed (Participants) | 3
  Change From Baseline at Completion/ termination (Month 36): 13-<16 years | 3.62 (5.471)
  Change From Baseline at End of Epoch 2: 2-4 years: number analyzed (Participants) | 8
  Change From Baseline at End of Epoch 2: 2-4 years | 8.16 (17.730)
  Change From Baseline at End of Epoch 2: 5-7 years: number analyzed (Participants) | 9
  Change From Baseline at End of Epoch 2: 5-7 years | -4.59 (16.266)
  Change From Baseline at End of Epoch 2: 8-12 years: number analyzed (Participants) | 17
  Change From Baseline at End of Epoch 2: 8-12 years | -1.98 (14.027)
  Change From Baseline at End of Epoch 2: 13-<16 years: number analyzed (Participants) | 8
  Change From Baseline at End of Epoch 2: 13-<16 years | -2.45 (8.807)

40. Secondary Outcome: HRQoL: Change From Baseline in EuroQol Five Dimensions Questionnaire (EQ-5D) Score
Description: The EQ-5D is a validated, self-administered assessment of overall health consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Participants were asked to describe their health state that day by choosing 1 of 3 responses that reflect the levels of severity for each of the five dimensions: no problems, some or moderate problems, or extreme problems. The domain scores are calculated with higher scores indicating worsening health status. The EQ-5D also includes a standard vertical 20-cm visual analogue scale (similar to a thermometer) for recording a participant's rating of their current HRQoL state, which ranged from 0 to 100, where 0 indicated worst imaginable health state and 100 was best imaginable health state. End of Epoch 2 summarizes all participant's data for their last epoch 2 visit (so not including the participant that discontinued in epoch 1).
Time Frame: Epoch 1: Baseline (First Infusion); Study Epoch 2: Up to Month 36
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epoch 1 + Epoch 2
Number analyzed (Participants) | 43
score on a scale
  Baseline: Visual Analogue Scale (VAS) Score | 82.84 (16.806)
  Baseline: Mobility | 1.07 (0.258)
  Baseline: Self-care | 1.16 (0.485)
  Baseline: Usual Activities | 1.14 (0.413)
  Baseline: Pain/ Discomfort | 1.28 (0.454)
  Baseline: Anxiety/ Depression | 1.28 (0.549)
  Change From Baseline at Epoch 2 Month 12: VAS Score: number analyzed (Participants) | 33
  Change From Baseline at Epoch 2 Month 12: VAS Score | 0.64 (23.504)
  Change From Baseline at Epoch 2 Month 12: Mobility: number analyzed (Participants) | 33
  Change From Baseline at Epoch 2 Month 12: Mobility | -0.09 (0.292)
  Change From Baseline at Epoch 2 Month 12: Self-care: number analyzed (Participants) | 33
  Change From Baseline at Epoch 2 Month 12: Self-care | -0.12 (0.415)
  Change From Baseline at Epoch 2 Month 12: Usual Activities: number analyzed (Participants) | 33
  Change From Baseline at Epoch 2 Month 12: Usual Activities | 0.03 (0.394)
  Change From Baseline at Epoch 2 Month 12: Pain/ Discomfort: number analyzed (Participants) | 33
  Change From Baseline at Epoch 2 Month 12: Pain/ Discomfort | 0.18 (0.528)
  Change From Baseline at Epoch 2 Month 12: Anxiety/ Depression: number analyzed (Participants) | 33
  Change From Baseline at Epoch 2 Month 12: Anxiety/ Depression | -0.06 (0.556)
  Change From Baseline at Completion/ Termination (Month 36): VAS Score: number analyzed (Participants) | 15
  Change From Baseline at Completion/ Termination (Month 36): VAS Score | -8.93 (26.993)
  Change From Baseline at Completion/ Termination (Month 36): Mobility: number analyzed (Participants) | 15
  Change From Baseline at Completion/ Termination (Month 36): Mobility | 0.00 (0.000)
  Change From Baseline at Completion/ Termination (Month 36): Self-care: number analyzed (Participants) | 15
  Change From Baseline at Completion/ Termination (Month 36): Self-care | 0.00 (0.000)
  Change From Baseline at Completion/ Termination (Month 36): Usual Activities: number analyzed (Participants) | 15
  Change From Baseline at Completion/ Termination (Month 36): Usual Activities | 0.00 (0.535)
  Change From Baseline at Completion/ Termination (Month 36): Pain/ Discomfort: number analyzed (Participants) | 15
  Change From Baseline at Completion/ Termination (Month 36): Pain/ Discomfort | -0.07 (0.594)
  Change From Baseline at Completion/ Termination (Month 36): Anxiety/ Depression: number analyzed (Participants) | 15
  Change From Baseline at Completion/ Termination (Month 36): Anxiety/ Depression | -0.27 (0.594)
  Change From Baseline at End of Epoch 2: VAS Score: number analyzed (Participants) | 41
  Change From Baseline at End of Epoch 2: VAS Score | -2.83 (24.895)
  Change From Baseline at End of Epoch 2: Mobility: number analyzed (Participants) | 41
  Change From Baseline at End of Epoch 2: Mobility | -0.07 (0.264)
  Change From Baseline at End of Epoch 2: Self-care: number analyzed (Participants) | 41
  Change From Baseline at End of Epoch 2: Self-care | -0.10 (0.374)
  Change From Baseline at End of Epoch 2: Usual Activities: number analyzed (Participants) | 41
  Change From Baseline at End of Epoch 2: Usual Activities | 0.00 (0.387)
  Change From Baseline at End of Epoch 2: Pain/ Discomfort: number analyzed (Participants) | 41
  Change From Baseline at End of Epoch 2: Pain/ Discomfort | 0.07 (0.565)
  Change From Baseline at End of Epoch 2: Anxiety/ Depression: number analyzed (Participants) | 41
  Change From Baseline at End of Epoch 2: Anxiety/ Depression | -0.10 (0.539)

41. Secondary Outcome: Treatment Preference and Satisfaction: Change From Baseline in Assessment of Life Quality Index (LQI) Score
Description: The LQI is a validated questionnaire assessing participant perceptions of their HRQoL and their treatment specifically among participants who use IgG therapy. This questionnaire covers 4 domains: treatment interferences, therapy-related problems, therapy setting, and treatment costs. The LQI domains are scored from 0 to 100, with higher scores associated with better IgG treatment satisfaction. End of Epoch 2 summarizes all participant's data for their last epoch 2 visit (so not including the participant that discontinued in epoch 1).
Time Frame: Epoch 1: Baseline (First Infusion); Study Epoch 2: Up to Month 36
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epoch 1 + Epoch 2
Number analyzed (Participants) | 43
score on a scale
  Baseline: Treatment Interferences | 69.77 (17.518)
  Baseline: Therapy-related Problems | 65.21 (17.080)
  Baseline: Therapy Setting | 85.66 (14.610)
  Baseline: Treatment Costs | 60.85 (27.310)
  Change From Baseline at Epoch 2 Month 12: Treatment Interferences: number analyzed (Participants) | 33
  Change From Baseline at Epoch 2 Month 12: Treatment Interferences | 4.71 (18.419)
  Change From Baseline at Epoch 2 Month 12: Therapy-related Problems: number analyzed (Participants) | 33
  Change From Baseline at Epoch 2 Month 12: Therapy-related Problems | 4.67 (17.670)
  Change From Baseline at Epoch 2 Month 12: Therapy Setting: number analyzed (Participants) | 33
  Change From Baseline at Epoch 2 Month 12: Therapy Setting | -6.23 (23.189)
  Change From Baseline at Epoch 2 Month 12: Treatment Costs: number analyzed (Participants) | 33
  Change From Baseline at Epoch 2 Month 12: Treatment Costs | 4.55 (36.330)
  Change From Baseline at Completion/Termination (Month 36): Treatment Interferences: number analyzed (Participants) | 14
  Change From Baseline at Completion/Termination (Month 36): Treatment Interferences | -10.52 (23.850)
  Change From Baseline at Completion/Termination (Month 36): Therapy-related Problems: number analyzed (Participants) | 14
  Change From Baseline at Completion/Termination (Month 36): Therapy-related Problems | -13.39 (31.656)
  Change From Baseline at Completion/Termination (Month 36): Therapy Setting: number analyzed (Participants) | 14
  Change From Baseline at Completion/Termination (Month 36): Therapy Setting | -15.87 (27.808)
  Change From Baseline at Completion/Termination (Month 36): Treatment Costs: number analyzed (Participants) | 14
  Change From Baseline at Completion/Termination (Month 36): Treatment Costs | -1.19 (32.826)
  Change From Baseline at End of Epoch 2: Treatment Interferences: number analyzed (Participants) | 41
  Change From Baseline at End of Epoch 2: Treatment Interferences | 1.49 (20.908)
  Change From Baseline at End of Epoch 2: Therapy-related Problems: number analyzed (Participants) | 41
  Change From Baseline at End of Epoch 2: Therapy-related Problems | 0.41 (24.399)
  Change From Baseline at End of Epoch 2: Therapy Setting: number analyzed (Participants) | 41
  Change From Baseline at End of Epoch 2: Therapy Setting | -10.16 (24.718)
  Change From Baseline at End of Epoch 2: Treatment Costs: number analyzed (Participants) | 41
  Change From Baseline at End of Epoch 2: Treatment Costs | 4.27 (35.164)

42. Secondary Outcome: Treatment Preference and Satisfaction: Change From Baseline in Assessment of Treatment Satisfaction and Medication Questionnaire (TSQM-9) Score
Description: The TSQM-9 is a 9-item, validated, self-administered instrument to assess participant satisfaction with medication, which assesses 3 domains: effectiveness, convenience, and global satisfaction. The TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction. End of Epoch 2 summarizes all participant's data for their last epoch 2 visit (so not including the participant that discontinued in epoch 1).
Time Frame: Epoch 1: Baseline (First Infusion); Study Epoch 2: Up to Month 36
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Epoch 1 + Epoch 2
Number analyzed (Participants) | 43
score on a scale
  Baseline: Effectiveness | 74.81 (15.494)
  Baseline: Convenience | 66.15 (16.436)
  Baseline: Global Satisfaction | 79.07 (16.525)
  Change From Baseline at Epoch 2, Month 12: Effectiveness: number analyzed (Participants) | 33
  Change From Baseline at Epoch 2, Month 12: Effectiveness | 6.40 (16.204)
  Change From Baseline at Epoch 2, Month 12: Convenience: number analyzed (Participants) | 33
  Change From Baseline at Epoch 2, Month 12: Convenience | 2.19 (19.834)
  Change From Baseline at Epoch 2, Month 12: Global Satisfaction: number analyzed (Participants) | 33
  Change From Baseline at Epoch 2, Month 12: Global Satisfaction | 4.76 (18.529)
  Change From Baseline at Completion/ termination (Month 36): Effectiveness: number analyzed (Participants) | 14
  Change From Baseline at Completion/ termination (Month 36): Effectiveness | -12.70 (33.577)
  Change From Baseline at Completion/ termination (Month 36): Convenience: number analyzed (Participants) | 14
  Change From Baseline at Completion/ termination (Month 36): Convenience | -7.14 (20.375)
  Change From Baseline at Completion/ termination (Month 36): Global Satisfaction: number analyzed (Participants) | 14
  Change From Baseline at Completion/ termination (Month 36): Global Satisfaction | -17.35 (36.283)
  Change From Baseline at end of Epoch 2: Effectiveness: number analyzed (Participants) | 41
  Change From Baseline at end of Epoch 2: Effectiveness | 3.52 (20.591)
  Change From Baseline at end of Epoch 2: Convenience: number analyzed (Participants) | 41
  Change From Baseline at end of Epoch 2: Convenience | -0.81 (20.244)
  Change From Baseline at end of Epoch 2: Global Satisfaction: number analyzed (Participants) | 41
  Change From Baseline at end of Epoch 2: Global Satisfaction | -0.17 (24.406)

43. Secondary Outcome: Treatment Preference and Satisfaction: Number of Participants Who Completed Treatment Preference Questionnaire
Description: The treatment preference questionnaire, internally developed by the study sponsor, is a self-administered, non-validated scale assessing participant preference for various attributes of immunoglobulin G (IgG) therapy.End of Epoch 2 summarizes all participant's data for their last epoch 2 visit (so not including the participant that discontinued in epoch 1).
Time Frame: Study Epoch 2: Up to Month 36
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Epoch 2
Number analyzed (Participants) | 43
Participants
  Month 12 | 34
  Completion/ Termination (Month 36) | 14
  End of Epoch 2 | 42

44. Secondary Outcome: Health Resource Utilization: Days Not Able to go to School or Work, or to Perform Normal Daily Activities
Description: Days not able to go to school or work, or to perform normal daily activities due to infection or other illnesses were calculated as days not able to go to school or work, or to perform normal daily activities due to infection or other illnesses per participant-year. Per participant-years = number or days reported / total number of years of study duration, i.e., the sum of study duration for all participants in the analysis set, divided by 365.25.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Number; unit: days per participant-year
Units Other Than Participants: Years
Arm/Group | Epoch 1 + Epoch 2
Number analyzed (Participants) | 44
Number analyzed (Years) | 52
days per participant-year | 4.28

45. Secondary Outcome: Health Resource Utilization: Days on Antibiotics
Description: Days on antibiotics were calculated as days on antibiotics per participant-year. Per participant-years = number or days reported / total number of years of study duration, i.e., the sum of study duration for all participants in the analysis set, divided by 365.25.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Number; unit: days per participant-year
Units Other Than Participants: Infusion
Arm/Group | Epoch 1 + Epoch 2
Number analyzed (Participants) | 44
Number analyzed (Infusion) | 52
days per participant-year | 26.77

46. Secondary Outcome: Health Resource Utilization: Number of Hospitalizations
Description: Number of hospitalizations, indication for the hospitalization (infection or non-infection) were calculated as number of hospitalizations, indication for the hospitalization (infection or non-infection) per participant-year. Per participant-years = number or days reported / total number of years of study duration, i.e., the sum of study duration for all participants in the analysis set, divided by 365.25.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Number; unit: hospitalizations per participant-year
Arm/Group | Epoch 1 + Epoch 2
Number analyzed (Participants) | 44
hospitalizations per participant-year | 0.08

47. Secondary Outcome: Health Resource Utilization: Number of Days Hospitalized Per Participant-Year
Description: Number of days hospitalized were calculated as number of days hospitalized per participant-year. Per participant-years = number or days reported / total number of years of study duration, i.e., the sum of study duration for all participants in the analysis set, divided by 365.25.
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Population: SAS included all participants who received at least one dose of HyQvia.
Measure: Number; unit: days per participant-year
Units Other Than Participants: Participant-Years
Arm/Group | Epoch 1 + Epoch 2
Number analyzed (Participants) | 44
Number analyzed (Participant-Years) | 52
days per participant-year | 0.21

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to EOS (up to 4 years 9 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant via the participant diary or observed by the investigator was recorded, irrespective of the relation to study treatment. SAS included all participants who received at least one dose of HYQVIA.
Arm/Group | Epoch 1 | Epoch 2
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/44 | 3/43
Other Adverse Events (participants affected / at risk) | 28/44 | 40/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epoch 1 (N=44) | Epoch 2 (N=43)
Adenovirus infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoch 1 (N=44) | Epoch 2 (N=43)
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Acute sinusitis (Infections and infestations) | 0 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bronchitis (Infections and infestations) | 0 | 3
Chills (General disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 5
Dizziness (Nervous system disorders) | 0 | 4
Ear infection (Infections and infestations) | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Fatigue (General disorders) | 5 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 3
Headache (Nervous system disorders) | 7 | 16
Influenza (Infections and infestations) | 0 | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 4
Infusion site erythema (General disorders) | 5 | 10
Infusion site extravasation (General disorders) | 2 | 10
Infusion site pain (General disorders) | 10 | 15
Infusion site pruritus (General disorders) | 3 | 10
Infusion site swelling (General disorders) | 3 | 9
Injection site pain (General disorders) | 7 | 1
Nausea (Gastrointestinal disorders) | 2 | 6
Otitis externa (Infections and infestations) | 0 | 3
Otitis media (Infections and infestations) | 2 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Pharyngitis (Infections and infestations) | 0 | 3
Pharyngitis streptococcal (Infections and infestations) | 1 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5
Pyrexia (General disorders) | 0 | 12
Rash (Skin and subcutaneous tissue disorders) | 0 | 5
Sinusitis (Infections and infestations) | 4 | 16
Upper respiratory tract infection (Infections and infestations) | 1 | 8
Viral upper respiratory tract infection (Infections and infestations) | 2 | 8
Vomiting (Gastrointestinal disorders) | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT03277313/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT03277313/SAP_001.pdf